CLINICAL TRIAL: NCT00006297
Title: Risk Factors for CV Disease in a Dialysis Cohort
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 914; R01HL062985 (NIH)
Record Dates: First submitted 2000-09-25; First posted 2000-09-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Kidney Failure, Chronic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Kidney Failure, Chronic

SUMMARY:
To investigate whether traditional risk factors and novel risk factors predict higher risk of atherosclerotic cardiovascular disease (ASCVD) in a prospective study of incident dialysis patients.

DETAILED DESCRIPTION:
BACKGROUND:

There is a very high mortality especially from cardiovascular disease among patients who are on dialysis. Atherosclerotic cardiovascular disease (ASCVD) is a leading contributor to the high morbidity and mortality among end-stage renal disease (ESRD) patients, accounting for 36 percent of ESRD deaths (total annual mortality of 23 percent). The high mortality among dialysis patients is a major public health problem and the ability to identify and treat risk factors that may reduce morbidity and mortality would be of substantial benefit. There are well-known risk factors for cardiovascular disease that certainly are related to morbidity and mortality among dialysis patients, i.e., relationship to hypertension, diabetes, smoking, etc. However, some of the new risk factors could also contribute to the excess mortality.

DESIGN NARRATIVE:

The prospective study tested the hypothesis that higher levels of several novel risk factors (Lp(a) levels and apo(a) isoforms; homocysteine and related vitamins; Chlamydia pneumoniae and cytomegalovirus; and C-reactive protein and fibrinogen) and traditional risk factors predicted higher risk of ASCVD in 925 incident dialysis patients recruited within three months of starting dialysis. Although these factors had been implicated in the etiology of ASCVD in ESRD patients, little prospective data existed. The cohort had already been recruited through a collaboration between Johns Hopkins and 80 Dialysis Clinics Incorporated (DCI) clinics; many of the important predictors and possible confounders had been measured. Long-term follow-up was obtained by extending mean followup of 2.4 years by four more years.

The investigators 1) extended specimen collection, and follow-up, and instituted standardized review of ASCVD events; 2) characterized baseline associations of novel and traditional factors with each other, dialysis modality and dose, nutritional status, and ASCVD prevalence in the full cohort using a cross-sectional design; 3) determined whether baseline levels of risk factors predicted subsequent incidence of ASCVD events, and total mortality using a prospective cohort study design and tested a priori hypothesized interactions between risk factors and the risk of ASCVD; 4) studied the variability of risk factors over time using annual measurements in a random subset of 180 patients (subcohort) using a longitudinal design; and lastly, 5) used a case-cohort design, utilizing the subcohort, to test whether the most recent level before an ASCVD event, the baseline level, or the mean level of each risk factor was most predictive of ASCVD risk. Baseline data collection included a patient health questionnaire and a standardized review of comorbidity using dialysis chart records. Serum, plasma and DNA were stored at -80 degrees C. from patient visits at recruitment (month 0), and followup (months 1,2,3,6,12,8,24, etc.). ASCVD was assessed by review of hospital charts, patients and care providers questionnaires, and HCFA death forms.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Coresh — Johns Hopkins University

REFERENCES:
- [Background] Miskulin DC, Meyer KB, Martin AA, Fink NE, Coresh J, Powe NR, Klag MJ, Levey AS; Choices for Healthy Outcomes in Caring for End-Stage Renal Disease (CHOICE) Study. Comorbidity and its change predict survival in incident dialysis patients. Am J Kidney Dis. 2003 Jan;41(1):149-61. doi: 10.1053/ajkd.2003.50034. PMID 12500232
- [Background] Astor BC, Eustace JA, Klag MJ, Powe NR, Longenecker JC, Fink NE, Marcovina SM, Coresh J; CHOICE Study. Race-specific association of lipoprotein(a) with vascular access interventions in hemodialysis patients: the CHOICE Study. Kidney Int. 2002 Mar;61(3):1115-23. doi: 10.1046/j.1523-1755.2002.00194.x. PMID 11849466
- [Background] Astor BC, Eustace JA, Powe NR, Klag MJ, Sadler JH, Fink NE, Coresh J. Timing of nephrologist referral and arteriovenous access use: the CHOICE Study. Am J Kidney Dis. 2001 Sep;38(3):494-501. doi: 10.1053/ajkd.2001.26833. PMID 11532680
- [Background] Liu Y, Coresh J, Eustace JA, Longenecker JC, Jaar B, Fink NE, Tracy RP, Powe NR, Klag MJ. Association between cholesterol level and mortality in dialysis patients: role of inflammation and malnutrition. JAMA. 2004 Jan 28;291(4):451-9. doi: 10.1001/jama.291.4.451. PMID 14747502
- [Background] Plantinga LC, Fink NE, Sadler JH, Levey AS, Levin NW, Rubin HR, Coresh J, Klag MJ, Powe NR. Frequency of patient-physician contact and patient outcomes in hemodialysis care. J Am Soc Nephrol. 2004 Jan;15(1):210-8. doi: 10.1097/01.asn.0000106101.48237.9d. PMID 14694175
- [Background] Longenecker JC, Coresh J, Marcovina SM, Powe NR, Levey AS, Giaculli F, Fink NE, Klag MJ. Lipoprotein(a) and prevalent cardiovascular disease in a dialysis population: The Choices for Healthy Outcomes in Caring for ESRD (CHOICE) study. Am J Kidney Dis. 2003 Jul;42(1):108-16. doi: 10.1016/s0272-6386(03)00413-x. PMID 12830462
- [Background] Fox CS, Longenecker JC, Powe NR, Klag MJ, Fink NE, Parekh R, Coresh J; CHOICE Study. Undertreatment of hyperlipidemia in a cohort of United States kidney dialysis patients. Clin Nephrol. 2004 May;61(5):299-307. doi: 10.5414/cnp61299. PMID 15182124
- [Background] Unruh ML, Levey AS, D'Ambrosio C, Fink NE, Powe NR, Meyer KB; Choices for Healthy Outcomes in Caring for End-Stage Renal Disease (CHOICE) Study. Restless legs symptoms among incident dialysis patients: association with lower quality of life and shorter survival. Am J Kidney Dis. 2004 May;43(5):900-9. doi: 10.1053/j.ajkd.2004.01.013. PMID 15112181
- [Background] Plantinga LC, Fink NE, Jaar BG, Sadler JH, Coresh J, Klag MJ, Levey AS, Powe NR. Frequency of sit-down patient care rounds, attainment of clinical performance targets, hospitalization, and mortality in hemodialysis patients. J Am Soc Nephrol. 2004 Dec;15(12):3144-53. doi: 10.1097/01.ASN.0000146424.91128.2A. PMID 15579518
- [Background] Jaar BG, Coresh J, Plantinga LC, Fink NE, Klag MJ, Levey AS, Levin NW, Sadler JH, Kliger A, Powe NR. Comparing the risk for death with peritoneal dialysis and hemodialysis in a national cohort of patients with chronic kidney disease. Ann Intern Med. 2005 Aug 2;143(3):174-83. doi: 10.7326/0003-4819-143-3-200508020-00003. PMID 16061915
- [Background] Liu Y, Berthier-Schaad Y, Fink NE, Fallin MD, Tracy RP, Klag MJ, Smith MW, Coresh J. Beta-fibrinogen haplotypes and the risk for cardiovascular disease in a dialysis cohort. Am J Kidney Dis. 2005 Jul;46(1):78-85. doi: 10.1053/j.ajkd.2005.03.008. PMID 15983960
- [Background] Longenecker JC, Klag MJ, Marcovina SM, Liu YM, Jaar BG, Powe NR, Fink NE, Levey AS, Coresh J. High lipoprotein(a) levels and small apolipoprotein(a) size prospectively predict cardiovascular events in dialysis patients. J Am Soc Nephrol. 2005 Jun;16(6):1794-802. doi: 10.1681/ASN.2004110922. Epub 2005 Mar 30. PMID 15800123
- [Background] Astor BC, Eustace JA, Powe NR, Klag MJ, Fink NE, Coresh J; CHOICE Study. Type of vascular access and survival among incident hemodialysis patients: the Choices for Healthy Outcomes in Caring for ESRD (CHOICE) Study. J Am Soc Nephrol. 2005 May;16(5):1449-55. doi: 10.1681/ASN.2004090748. Epub 2005 Mar 23. PMID 15788468
- [Background] Plantinga LC, Jaar BG, Fink NE, Sadler JH, Levin NW, Coresh J, Klag MJ, Powe NR. Frequency of patient-physician contact in chronic kidney disease care and achievement of clinical performance targets. Int J Qual Health Care. 2005 Apr;17(2):115-21. doi: 10.1093/intqhc/mzi010. Epub 2005 Feb 21. PMID 15723821